CLINICAL TRIAL: NCT06572189
Title: The Safety and Efficacy of Transarterial Injection of CD-801 in Patients With Advanced Intrahepatic Cholangiocarcinoma
Brief Title: The Safety and Efficacy of CD-801 in Patients With Advanced Intrahepatic Cholangiocarcinoma
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Based on the results of another intravenous injection therapy CD-801 for the treatment of hepatocellular carcinoma, we have decided to change the administration method and therefore withdraw this trial protocol.
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Wei-Fen Xie, Professor, Shanghai Changzheng Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024SL015
Record Dates: First submitted 2024-08-06; First posted 2024-08-27 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Intrahepatic Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD-801, a lipid nanoparticle-encapsulated self-replicating RNA encoding hepatocyte nuclear factor 4α (Experimental): Patients will receive administration of 100μg of CD-801 via hepatic arterial injection every 14 ± 3 days
  Interventions: Genetic: Injection of CD-801, a lipid nanoparticle-encapsulated self-replicating RNA encoding hepatocyte nuclear factor 4α (HNF4α)

INTERVENTIONS:
Genetic: Injection of CD-801, a lipid nanoparticle-encapsulated self-replicating RNA encoding hepatocyte nuclear factor 4α (HNF4α) — Receive administration of 100μg of CD-801 via hepatic arterial injection every 14 ± 3 days (the dosing interval will be adjusted based on the tolerability, safety, and therapeutic effect of the subjects), for one treatment cycle. Treatment will continue until the occurrence of disease progression, death, intolerable toxicity, voluntary withdrawal of informed consent, loss to follow-up, initiation of new antitumor treatment, or termination of the study by the investigator (whichever comes first), and completion of the final follow-up and assessment 14 days after the last administration.

SUMMARY:
The goal of this clinical trial is to learn about the safety of CD-801, a lipid nanoparticle-encapsulated self-replicating RNA encoding hepatocyte nuclear factor 4α (HNF4α) in treating patients with advanced intrahepatic cholangiocarcinoma (ICC). It will also learn if CD-801 works to treat advanced ICC. The main questions it aims to answer are:

1. What medical problems do participants have when injecting CD-801?
2. Is CD-801 effective for ICC patients according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 or modified RECIST (mRECIST)

Participants will:

Receive administration of 100μg of CD-801 via hepatic arterial injection every 14 ± 3 days (the dosing interval will be adjusted based on the tolerability, safety, and therapeutic effect of the subjects), for one treatment cycle. Treatment will continue until the occurrence of disease progression, death, intolerable toxicity, voluntary withdrawal of informed consent, loss to follow-up, initiation of new antitumor treatment, or termination of the study by the investigator (whichever comes first), and completion of the final follow-up and assessment 14 days after the last administration.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, aged 18 years or older.
* Histologically or cytologically confirmed intrahepatic cholangiocarcinoma patients.
* Patients with intrahepatic cholangiocarcinoma not suitable for surgical resection, liver transplantation, or ablation therapy, or those with post-surgical recurrence and/or metastasis.
* Patients not suitable for local or systemic treatment, or those who have progressed after at least one chemotherapy regimen containing gemcitabine/fluoropyrimidine/platinum, etc..
* Life expectancy of 12 weeks or more.
* Subjects must have an Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 to 2.
* Males with fertility and females of childbearing potential are willing to use a highly effective method of contraception for the entire study period and for 6 months after study drug discontinuation. Females of childbearing age, including premenopausal females and within 2 years after menopause, must have a negative serum pregnancy test result within 7 days prior to the first dose of study treatment.
* Subjects who had a voluntary agreement to provide written informed consent and the willingness and ability to comply with all aspects of the protocol.

Exclusion Criteria:

* Patients with any of the following criteria were excluded from participation in this study:

  * Inadequate liver function：Albumin (ALB) < 25 g/L, or total bilirubin > 5 × the upper limit of normal (ULN), or aspartate aminotransferase (AST), alkaline phosphatase (ALP), or alanine aminotransferase (ALT) >10 × ULN.
  * Inadequate renal function defined as creatinine >1.5 × ULN or calculated creatinine clearance < 40 mL/min.
  * Absolute neutrophil count (ANC) < 1.0×109/L, or Platelets < 30×109/L, or Hemoglobin < 8.5 g/dL.
  * International normalized ratio (INR) > 2.3.
  * Poorly controlled hypertension, diabetes or other serious heart or lung diseases, or with serious dysfunction.
  * Patients who have received local or systemic anti-tumor treatments such as ablation, Transhepatic Arterial Chemotherapy and Embolization (TACE), local radiotherapy of the liver, immunotherapy, targeted therapy, etc., within 4 weeks, or chemotherapy, other trial drugs, or radiotherapy of metastatic lesions within 2 weeks, except for treatment regimens assessed as disease progression according to mRECIST or RECIST 1.1.
  * Patients with uncurable brain metastasis.
  * All toxicities related to prior locoregional or systemic anti-tumor treatments are still grade 2 or more (except for hair loss and other events that have been judged tolerable by researchers).
  * Complication histories of liver cirrhosis or HCC such as gastrointestinal hemorrhage, overt hepatic encephalopathy, or refractory ascites within 2 weeks prior to the first dose of study treatment.
  * Uncontrolled active infection (eg, lung infections, or abdominal infections).
  * History of malignancy other than HCC within 5 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death (e.g., 5-year overall survival rate > 90%), such as adequately treated early gastric carcinoma, carcinoma in situ of the cervix, non-melanoma skin carcinoma, or localized prostate cancer.
  * Hepatitis B virus DNA greater than 500 copies/mL, or hepatitis C virus RNA greater than 15 U/mL.
  * Positive for human immunodeficiency virus (HIV).
  * Allergic to contrast agents.
  * Pregnant/lactating women, or women with the possibility of pregnancy.
  * Any medical conditions which, in the opinion of the investigator, would preclude participation in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-08-28 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | up to 24 months
  The incidence, timing, and severity of adverse events, serious adverse events, and adverse events leading to treatment discontinuation according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0.

SECONDARY OUTCOMES:
Objective Response Rate | up to 24 months
  The proportion of subjects achieving Complete Response (CR) and Partial Response (PR).
Duration Of Response | up to 24 months
  The time from the first documentation of response (either Partial Response or Complete Response) after the start of treatment to the first documentation of disease progression or death due to Intrahepatic Cholangiocarcinoma (ICC), whichever occurs first.
Progression-Free Survival | From date of the start of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  The time from the start of treatment to the first occurrence of disease progression or death due to Hepatocellular Carcinoma (HCC), whichever comes first.
  The time from the initiation of treatment to the first documentation of disease progression or death due to Intrahepatic Cholangiocarcinoma (ICC), whichever occurs first.
Time To Progression | up to 24 months
  The time from the start of treatment to the first recorded documentation of disease progression, excluding death.
Time To Response | up to 24 months
  The time from the commencement of treatment to the first documentation of response achieving either Partial Response (PR) or Complete Response (CR).
Disease Control Rate | up to 24 months
  The proportion of subjects achieving response with either Partial Response (PR) or Complete Response (CR), or maintaining stable disease (SD with duration of ≥ 5 weeks) after treatment.
Clinical Benefit Rate | up to 24 months
  The proportion of subjects who achieve either a Partial Response (PR) or Complete Response (CR) following treatment, or maintain durable stable disease (SD with a duration of at least 23 weeks).
Overall Survival | From date of the start of treatment until the date of death from any cause, assessed up to 36 months
  The time from the start of treatment to death from any cause.
Patient Reported Outcome-1 | up to 24 months
  the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30)
Patient Reported Outcome-2 | up to 24 months
  the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire BIL21 (QLQ-BIL21)
Patient Reported Outcome-3 | up to 24 months
  The Generic Euroquol Five Dimension Five Level (EQ-5D-5L) Questionnaire
The changes in tumor markers after treatment. | up to 24 months
  The changes in tumor markers such as CA19-9, Carcinoembryonic Antigen (CEA), and Alpha-fetoprotein (AFP) after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Wen-Ping Xu, Shanghai, Shanghai Municipality, China